CLINICAL TRIAL: NCT03345134
Title: Phase II Study of Pembrolizumab in Combination With BCG After Endoscopic Ablation for Patients With High Risk Superficial Upper Urinary Tract Transitional Cell Carcinoma Unfit or Unwilling to be Treated With Nephroureterectomy
Brief Title: Pembrolizumab in Combination With BCG After Ablation in Patients With UUTTCC Without Nephroureterectomy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shaheen Alanee (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Shaheen Alanee, Senior Staff Physician Department of Urology, Henry Ford Health System
Organization: Henry Ford Health System (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HFHS 16-01
Record Dates: First submitted 2017-11-03; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: High Risk Superficial Upper Urinary Tract Transitional Cell Carcinoma; Endoscopic Surgical Procedure; Transitional Epithelial Cells
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- MK-3475 and BCG (Experimental): Single treatment group of high risk superficial upper urinary tract transitional cell carcinoma; combination treatment with MK-3475 and BCG
  Interventions: Drug: MK-3475 and BCG

INTERVENTIONS:
Drug: MK-3475 and BCG — combination treatment with MK-3475 and BCG after endoscopic ablation

SUMMARY:
PURPOSE: This study is being conducted to test the safety of the study drug Pembrolizumab, also known as MK-3475, at different dose levels in combination with the current therapy, (BCG), for superficial upper urinary tract transitional cell carcinoma. We want to find out what effects, good and/or bad, it has on upper urinary transitional cell carcinoma OBJECTIVE: To determine the safety of administering MK-3475 at a fixed dose of 200 mg every three weeks in conjunction with intrapelvic BCG treatment in high risk superficial UUTTCC patients who are unfit or unwilling to be treated with radical nephroureterectomy.

STUDY DESIGN: Open-label, single center, Phase II, treatment trial TREATMENT: BCG- BCG treatment could be delivered both through a retrograde ureteral catheter placed under fluoroscopic control or through an antegrade nephrostomy tube placed by interventional radiology. Treatment will be once a week for 6 weeks. BCG treatment will begin on Day 1 of Week 7. Depending on patient's response, they may have additional treatments beyond the 6 scheduled, but they will be outside of the patient's participation in this study. Pembrolizumab will be given through an intravenous needle once every 21 days (one cycle) for a total of 6 cycles. It will take 30 minutes for the infusion of the study drug. Pembrolizumab will be given on Day 1 of weeks 1, 4, 7, 10, 13, and 16 while BCG will be given on Day 1 of weeks 7-12.

PROCEDURES: Following informed consent, prescreening and screening procedures will be performed, which will include medical history review, baseline chest x ray and EKG, ureteroscopy and pulmonary function tests for final eligibility status. Once subject is eligible, they will undergo physical exams (every 3 weeks), vital signs and weight (each study visit), adverse event monitoring (each study visit), ECGs (screening visit), bloodwork (at screening and then every 3 weeks), urinalysis at selected study visits, and concomitant medication review (each study visit), and questionnaires (selected study visits). After subject has completed week 19, they will have a study discontinuation visit, followed by a 30 day follow up visit. The subject will then be followed at 3, 6, 9, 12, 18 and 24 months post treatment where vital status will be determined as well as disease recurrence status. Ureteroscopy will be performed as standard of care but will be considered measures for efficacy. Biopsy will be performed as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial.
2. Be at least18 years of age on day of signing informed consent.
3. Have pathologically documented high grade UUTTCC (CIS, Ta, T1) that could be completely ablated with ureteroscopy or through antegrade percutaneous access.
4. Subject must also unwilling or unfit to undergo treatment with radical nephroureterectomy
5. Have provided tissue from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion. Tissue must be obtained from the most recent upper urinary tract biopsy.
6. Have a performance status of 0-1 on the ECOG Performance Scale (Appendix A).
7. Demonstrate adequate organ function, all screening labs should be performed within 28 days of treatment initiation.
8. Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female subjects of childbearing potential should be willing to use 2 methods of birth control or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.5.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
10. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
11. Patients who received prior systemic chemotherapy, targeted small molecule therapy, or radiation therapy for UUTTCC are allowed into the study as long as there is confirmed recurrence of the disease after previous treatment and the patient is unwilling or unfit to undergo radical surgery.

Exclusion Criteria:

1. Currently has active or progressive metastatic disease. (Chest X-ray, Computerized Tomography [CT] urogram or Magnetic Resonance Imaging [MRI], and urogram are allowed to ascertain the superficial nature of the disease when indicated, but not required. If urogram protocol is not available or contrast allergy/poor renal function precludes such imaging, then non-contrast CT or MRI of the abdomen/pelvis within 90 days of study entry will suffice.)
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has had a prior monoclonal antibody within 4 weeks before study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
4. Has had prior systemic chemotherapy, targeted small molecule therapy, or radiation therapy for UUTTCC.
5. If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
6. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, localized prostate cancer with no recurrence after curative surgery or radiation, or in situ cervical cancer that has undergone potentially curative therapy. Lower urinary tract transitional cell carcinoma is also allowable on study as high risk transitional cell carcinoma is commonly multifocal, and intraluminal BCG therapy is also used for treatment of lower urinary tract lesions in a manner similar to that of UUTTCC.
7. Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
8. Has history of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease, or active , non-infectious pneumonitis.
9. Has an active infection, including a concurrent febrile illness, requiring systemic therapy.
10. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
11. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
12. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 4 months after the last dose of trial treatment.
13. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways) including anti-CD40 and anti-OX40 antibodies.
14. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
15. Has known active Hepatitis B (e.g., HBs Ag reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
16. Has known active tuberculosis. Subjects will not be specifically tested for the study; however, subjects that are tested within 28 days of beginning study or while on study and test positive with the PPD test before treatment should have active tuberculosis ruled out before therapy begins for their superficial renal pelvis cancer.
17. Has received a live vaccine within 30 days prior to the first dose of trial treatment.
18. Has an active urinary tract infection, gross hematuria, or known broken mucosal barrier of the renal pelvis.
19. Less than 14 days post renal pelvis biopsy, TUR, or traumatic catheterization.
20. Evidence of muscle invasive renal pelvis cancer, or transitional cell carcinoma of the upper urinary tract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-11-30 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Complete Response per ureteroscopy and pathological confirmation of tissue biopsy | At 19 weeks

SECONDARY OUTCOMES:
Complete Response per ureteroscopy and pathological confirmation of tissue biopsy | Up to 24 months

OTHER OUTCOMES:
Progression Free Survival per ureteroscopy and pathological confirmation of tissue biopsy | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shaheen Alanee, MD, MPH, MBA, Detroit, Michigan, United States

REFERENCES:
- [Derived] Jamil ML, Deebajah M, Sood A, Alanee S. Combination of pembrolizumab and BCG treatment after endoscopic ablation of high-risk superficial upper urinary tract urothelial carcinoma in patients not candidates for radical nephroureterectomy: protocol for phase-II study. BMJ Open. 2019 Dec 3;9(12):e027066. doi: 10.1136/bmjopen-2018-027066. PMID 31796469